CLINICAL TRIAL: NCT01078168
Title: Changes of Cerebral Spinal Fluid APPSα Levels Under Oral Therapy With Acitretin 30 mg Daily in Patients With Mild to Moderate Alzheimer's Disease: a Multicenter Prospective Randomised Placebo-controlled Parallel-group Study
Brief Title: Alzheimer's Disease Acitretin Medication
Acronym: ADAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: K. Lieb (Other)
Collaborators: Alzheimer Forschungsinitiative e.V. (AFI) (Unknown)
Responsible Party: Sponsor-Investigator, K. Lieb, Herr Univ.-Prof. Dr. med. Andreas Fellgiebel, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADAM; 2009-011881-27 (EudraCT Number)
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-07

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Acitretin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acitretin (Active Comparator): oral, 30 mg per day, day 1-28
  Interventions: Drug: Acitretin
- Placebo (Placebo Comparator): oral, day 1-28
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acitretin — 30mg per day from Day 1 to Day 28
  Other Names: Neotigason, Acicutan
  Arms: Acitretin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The trials investigates the changes of cerebral spinal fluid (CSF) soluble alpha-secretase cleaved APP (APPsα) levels under oral therapy with acitretin 30mg daily in patients with mild to moderate Alzheimer's disease (AD).The present study aims to demonstrate an enhancement of the α-secretase activity by acitretin as measured by increased CSF APPSα levels in human AD. Second, the safety and tolerability of acitretin in AD patients should be proven.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate AD (NINCDS-ADRDA criteria)
* Mini-Mental State Examination (MMSE): 27-14 points
* Geriatric Depression Scale ≤ 14

Exclusion Criteria:

* hereditary cognitive impairment
* known history of brain injuries
* Insufficient German language skills
* actual treatment with other potential disease modifying drugs of AD
* multimorbidity or significant organ (esp. liver or renal) dysfunction
* evidence of Non-AD neurodegenerative disorder (e.g. Parkinson)
* contraindication to acitretin such as osteoporosis, hypoalbuminaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-03; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fellgiebel, PD Dr., Principal Investigator — Department of psychiatry and psychotherapy, University medical center of the Johannes Gutenberg-University Mainz, Germany
Locations (2):
- Germany (2):
  - Department of psychiatry and psychotherapy, University medical center of the Johannes Gutenberg-University Mainz, Mainz, Rhineland-Palatinate
  - Universität Rostock, Rostock

RESULTS

PARTICIPANT FLOW:
Recruitment Details: University Medical Centre of the Johannes Gutenberg University, Mainz, and University Medical Centre, Rostock, May 2010 to January 2013
Pre-assignment Details: neuropsychiatric testing, general exclusion of e.g. depression or severe diseases affecting the trial
Period: Overall Study
Arm/Group | Acitretin | Placebo
Started | 11 | 11
Completed | 11 | 10
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acitretin | Placebo | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (9.6) | 73 (3.8) | 69.33 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  Germany | 11 | 10 | 21
MMSE [Mean (Standard Deviation); unit: units on a scale] — MMSE: Mini-Mental State Examination; can be used to systematically and thoroughly assess mental status; range: 0-30; a score of 23 or lower is indicative of cognitive impairment
  units on a scale | 20.4 (4.2) | 23.9 (4.3) | 22.2 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Cerebrospinal Fluid (CSF) Soluble Alpha-clevaed Amyloid Precursor Protein (APPsα) Concentration at Visit 3 Compared to Baseline
Description: Values were assessed via Western blotting technique. Normalization was conducted using hSA levels of the individual samples.
Time Frame: baseline and 4 weeks (visit 3)
Population: All patients were included with successful punctation at V1 and V3. For one Acitretin-treated patient not punctation at V3 was obtained (resulting n of 10).
Measure: Mean (Standard Deviation); unit: fold change (Visit 3/background)
Arm/Group | Acitretin | Placebo
Number analyzed (Participants) | 10 | 10
fold change (Visit 3/background) | 1.251 (0.4528) | 0.8741 (0.2592)
Statistical Analysis 1: Comparison: Acitretin vs Placebo; Test type: Superiority or Other; p = 0.0347, t-test, 2 sided — threshold: p<0.05; Mean Difference (Final Values) = 0.3769, 95% CI 2-sided [0.03025 to 0.7235]

ADVERSE EVENTS:
Arm/Group | Acitretin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/10
Other Adverse Events (participants affected / at risk) | 8/11 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acitretin (N=11) | Placebo (N=10)
persistent diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — diagnostic workup because of persistent diarrhea required hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acitretin (N=11) | Placebo (N=10)
headache (General disorders) | 0 (0) | 1 (1)
migraine (General disorders) | 0 (0) | 1 (1)
syncope (General disorders) | 0 (0) | 1 (1)
light headedness (General disorders) | 0 (0) | 1 (1)
derailment of blood glucose (General disorders) | 0 (0) | 1 (1)
lowered glucose tolerance (General disorders) | 0 (0) | 1 (1)
aggressiveness (General disorders) | 0 (0) | 1 (1)
muscular pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
cataract surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
memory defect due to anaesthesia (Surgical and medical procedures) | 0 (0) | 1 (1)
gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
severe diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
post-punctual syndrome (Surgical and medical procedures) | 1 (1) | 0 (0)
exfoliation of callus (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
dry lips (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
dry eyes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
hypertensive crisis (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
gingivitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
backpain (General disorders) | 1 (1) | 0 (0)
dry mouth (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
infection due to insect sting (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes